CLINICAL TRIAL: NCT01342627
Title: Sorafenib in Elderly Patients With Metastatic Renal Cell Carcinoma (SERCC Study) Impact of Adverse Events Management in Elderly mRCC Patients Treated With Sorafenib
Brief Title: Sorafenib in Elderly Patients With Metastatic Renal Cell Carcinoma
Acronym: SERCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-019726-14
Record Dates: First submitted 2010-11-29; First posted 2011-04-27 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal Carcinoma; Metastatic; Sorafenib; Elderly
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Experimental): Sorafenib will be orally administered at a daily dose of 400 mg taken twice daily without food, at least one hour before or two hours after eating. Four weeks of treatments will be considered as a cycle. Each patient enrolled in the study will received medications for topical therapy. Dermatological medications will be provided free.
  In case of toxicities, dose reduction/interruption is permitted according to protocol.
  In case of disease progression Sorafenib administration will be discontinued.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be orally administered at a daily dose of 400 mg taken twice daily without food, at least one hour before or two hours after eating. Four weeks of treatments will be considered as a cycle. Each patient enrolled in the study will received medications for topical therapy. Dermatological medications will be provided free.
  In case of toxicities, dose reduction/interruption is permitted according to the protocol.
  In case of disease progression Sorafenib administration will be discontinued.
  Other Names: Nexavar

SUMMARY:
Study Design This is a multicenter, open label, first line phase II study in elderly (≥ 65 years old) metastatic Renal Cell Carcinoma (mRCC) patients not suitable for any other currently approved treatment (bevacizumab+INF, cytokines or sunitinib) except for sorafenib.

Each patient treated with sorafenib enrolled in the study will be trained to observe the management tool for skin care. A study period of 3 years was estimated as follows: an enrollment period of 24 months and a further follow-up period of 12 months.

Objectives of the trial Primary objective The primary aim of this trial is the evaluation of the efficacy of a patient education program in the reduction of Hand-Foot Skin Reaction (HFSR).

Secondary Objectives

TO assess:

* The frequency of dose discontinuation, interruption and reduction
* The incidence of any grade diarrhoea, and other adverse events
* The overall Response Rate according to the RECIST criteria.
* Progression free survival (PFR) in study population and comparison of PFS between age sub groups in the current study population

DETAILED DESCRIPTION:
Rationale of the present study For several decades, the systemic management of metastatic renal cell cancer (mRCC) was confined to the use of interferon (IFN) and interleukin-2 (IL-2). Recently, options for the medical management of mRCC have been improved through the introduction of agents targeting tumour angiogenesis or intracellular pathways mediating growth and proliferation. Among these agents are the small molecule inhibitors sorafenib (Nexavar), sunitinib (Sutent), temsirolimus (Torisel) and everolimus, and the monoclonal antibody bevacizumab (Avastin). All these targeted agents have been shown significantly to extend progression-free or overall survival or both when compared with placebo or IFN therapy in the treatment of mRCC.

Adverse events are commonly observed in clinical practice by using these small molecule inhibitors in mRCC patients. Concerning the use of bevacizumab the most commonly observed adverse events are hypertension, proteinuria, bleeding and thrombosis. For sunitinib the most frequent adverse events include hand-foot syndrome, stomatitis, diarrhea, fatigue, hypothyroidism and hypertension.

Most common adverse events with sorafenib are hand foot skin reaction (HFSR) rash, desquamation, fatigue, diarrhea, nausea, hypothyroidism and hypertension.Several studies and recommendations have been published in order to suggest how to manage sorafenib adverse reactions and in particular the HFSR.

The aim of this study is to evaluate if patients education programs for the prevention of dermatological events (HFSR, rash, desquamation) can reduce the onset these adverse events (all grades). The reduction of dermatological adverse effects would concomitantly limit the frequencies of sorafenib dose reduction and interruptions in mRCC patients not suitable for cytokines or anti-angiogenesis (bevacizumab or sunitinib) therapy as first line treatment.

Treatment Administration Sorafenib will be orally administered at a daily dose of 400 mg taken twice daily without food, at least one hour before or two hours after eating. Four weeks of treatments will be considered as a cycle. Each patient enrolled in the study will received medications for topical therapy. Dermatological medications will be provided free.

In case of toxicities, dose reduction/interruption is permitted according to the flow charts/dose modifications.

In case of disease progression, or unacceptable toxicities Sorafenib administration will be discontinued.

The patient will be considered "out of treatment" if Sorafenib intake is stopped for more than 30 consecutive days and the patient will be considered for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Nephrectomized, metastatic Clear Cell RCC patients not suitable for cytokines or anti-angiogenesis (bevacizumab or sunitinib) therapy as first line treatment
2. Age ≥ 65years
3. ECOG Performance Status of ≤ 2
4. MSKCC prognostic score, good or intermediate
5. Life expectancy of at least 12 weeks.
6. Subjects with at least one uni-dimensional (for RECIST) measurable lesion. Lesions must be measured by CT/MRI-scan.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of therapy:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Platelet count ≥ 100,000/μl
   * Total bilirubin ≤ 1.5 times the upper limit of normal
   * ALT and AST ≤ 2.5 x upper limit of normal (≤ 5 x upper limit of normal for patients with liver involvement of their cancer)
   * Alkaline phosphatase ≤ 4 x upper limit of normal
   * PT-INR/PT ≤ 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
   * Serum creatinine ≤ 1.5 x upper limit of normal.
8. Ability to take correctly oral drugs.
9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
10. Written Informed Consent
11. To be able to understand medical instruction and to fill in the patient's diary. If not, check if adequately supported by his/her family.

Exclusion Criteria:

1. Previous first line treatment for mRCC. No adjuvant or neoadjuvant treatments are allowed.
2. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
3. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring antiarrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
4. History of previous or present seizure disorder requiring medication (such as steroids or anti-epileptics), organ allograft, HIV infection or chronic hepatitis B or C
5. Active clinically serious infections (≥ grade 2 NCI-CTC version 3.0)
6. Patients undergoing renal dialysis
7. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
8. Patients with evidence or history of bleeding diathesis
9. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
10. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
11. Known allergy to sorafenib or one of its constituents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary aim of this trial is the evaluation of the efficacy of a patient education program in the reduction of HFSR | From enrollment in the study until 1 year
  The primary aim is to determine the efficacy of the patient education program in reducing the incidence of HFSR(all grades).The efficacy is measured in terms of percentage of HFSR-free.Simon's methods will be used to calculate sample size(Simon R,1989).Considering the optimal two-stage design for phase II,considering a difference p1-p0=20% and fixing error probabilities(alfa=0.05 and beta=0.20),the number of patients for the first step is 16.The trial will be terminated if less than 7 HFSR-free patients will be seen.Otherwise the accrual will continue up to a total of 46 patients.

SECONDARY OUTCOMES:
Frequency of dose discontinuation, interruption and reduction | From enrollment in the study until 1 year
  Frequency of dose discontinuation, interruption and reduction
Incidence of any grade diarrhoea, and other adverse events | From enrollment in the study until 1 year
  Incidence of any grade diarrhoea, and other adverse events
Overall Response Rate | From enrollment in the study until 1 year
  Overall Response Rate according to the RECIST criteria
Progression free survival (PFR) | From enrollment in the study until 1 year
  Progression free survival (PFR) in study population and comparison of Progression Free Survival (PFS) between age sub groups in the current study population

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Fratino, oncologist, Principal Investigator — Centro di Riferimento Oncologico - IRCCS - Aviano
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Pordenone, Italy

REFERENCES:
- See also: web site of Centro di Riferimento Oncologico (sponsor and coordinator center) — http://www.cro.sanita.fvg.it/